CLINICAL TRIAL: NCT06548646
Title: Ultrasound-guided Thoracic Interfascial Plane Nerve Block Versus Erector Spinae Plane Block for Postoperative Pain Control in Patients Undergoing Modified Radical Mastectomy
Brief Title: Ultrasound-guided Thoracic Interfascial Plane Nerve Block Versus Erector Spinae Plane Block for Pain Control After Modified Radical Mastectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Safie ramez tewfeik abd el moneim (Other)
Responsible Party: Sponsor-Investigator, Safie ramez tewfeik abd el moneim, Dr, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MD178/2023
Record Dates: First submitted 2024-08-04; First posted 2024-08-12 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Postoperative Pain Following Modified Radical Mastectomy for Breast Cancer
Keywords: breast cancer; Modified Radical Mastectomy; Mastectomy; postoperative pain; Erector Spinae Plane Block; Thoracic Interfascial Plane Block
MeSH Terms: conditions — Breast Neoplasms; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: All clinical staff, including surgeons, and anesthetists except the one giving the block, nurses, investigators, and patients will be blinded to the treatment group assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thoracic Interfascial Plane Block (Experimental): the Thoracic Interfascial Plane Block, which includes Pecto-Intercostal Fascial Plane Block and Serratus Intercostal Fascial Plane Block, is a peripheral nerve block that targets the intercostal nerve branches scattered throughout the chest and axilla
  Interventions: Procedure: Thoracic Interfascial Plane Block
- Erector Spinae Plane Block (Active Comparator): Erector Spinae Plane Block (ESPB) is an anesthesia technique for providing effective analgesia during and after breast and abdominal surgery
  Interventions: Procedure: Erector Spinae Plane Block

INTERVENTIONS:
Procedure: Thoracic Interfascial Plane Block — The Thoracic Interfascial Plane Block (TIPB) is a regional anesthesia technique used to manage postoperative pain, particularly in thoracic and breast surgeries. This block involves the injection of a local anesthetic into the fascial plane between the thoracic muscles, targeting the nerves that supply the chest wall and upper abdominal area. It includes Pecto-Intercostal Fascial Plane Block (PIFB) and Serratus Intercostal Fascial Plane Block (SIFB).
  Other Names: Thoracic Nerve Block; TIPB
  Arms: Thoracic Interfascial Plane Block
Procedure: Erector Spinae Plane Block — The Erector Spinae Plane Block (ESPB) is a regional anesthesia technique used to manage pain, particularly in thoracic and abdominal surgeries. This block involves the injection of a local anesthetic into the plane between the erector spinae muscle and the transverse processes of the vertebrae.
  Other Names: ESPB
  Arms: Erector Spinae Plane Block

SUMMARY:
This study compares two methods of local pain control in patients undergoing Modified Radical Mastectomy, a common surgery for breast cancer( tumor in the breast) treatment. It aims to determine which method, the Thoracic Interfascial Plane Block or the Erector Spinae Plane Block, provides better pain relief after surgery, reduces side effects, and increases patient satisfaction.

Why This Study Is Important:

Breast cancer surgery can cause significant pain, and managing this pain is important for a quick recovery. Currently, pain is often managed with opioids, which can cause side effects like nausea and drowsiness. invistigators want to find a method that controls pain effectively with fewer side effects, helping patients recover faster and feel better.

Who Can Take Part:

Women aged 21 and older who are scheduled for a Modified Radical Mastectomy at Ain Shams University hospitals can participate in this study.

What Will Happen During the Study:

Participants will be randomly assigned to receive either the Thoracic Interfascial Plane Block or the Erector Spinae Plane Block before surgery.

Pain levels will be measured using a numerical pain score from 1 to 10. Researchers will track the amount of pain medication needed, the time it takes to feel pain relief, and any side effects.

Other factors such as sleep quality, time to start walking again, and overall satisfaction with pain control will also be recorded.

What investigators hope to Learn:

Investigators hope to find out which nerve block provides better pain relief after surgery. By comparing TIPB and ESPB, with the aim to identify the method that:

Requires less additional pain medication Has fewer side effects Improves sleep quality and overall recovery Increases patient satisfaction

Significance:

This study could lead to better pain management strategies for breast cancer surgery, reducing the need for opioids and enhancing patient recovery and comfort.

Participation:

Participants will be monitored closely during and after the procedure to ensure their safety and well-being. The results of this study could help improve pain management for future patients undergoing similar surgeries.

DETAILED DESCRIPTION:
This study is a randomized, double-blinded clinical trial comparing the efficacy of two ultrasound-guided nerve blocks for postoperative pain management in patients undergoing Modified Radical Mastectomy (MRM). The two techniques under investigation are the Thoracic Interfascial Plane Block (TIPB) and the Erector Spinae Plane Block (ESPB). Both nerve blocks are administered to provide targeted pain relief by numbing specific nerves involved in the surgical area.

Methodology:

Participants will be randomly assigned to one of two groups to receive either TIPB or ESPB. The randomization will ensure unbiased distribution of participants across both groups. The nerve blocks will be administered preoperatively under ultrasound guidance to ensure accurate placement and effectiveness.

Assessments and Measurements:

Pain levels will be assessed using the Visual Analog Scale (VAS) at multiple time points postoperatively, including at rest and during movement. The primary outcome measure is the total amount of rescue pain medication required within the first 48 hours after surgery. Secondary outcomes include the time to first rescue analgesic, intraoperative fentanyl consumption, hemodynamic parameters, sleep quality, time to first ambulation, VAS scores for pain and nausea, and overall patient satisfaction.

Safety and Monitoring:

Participants will be monitored for adverse events, including complications related to the nerve block techniques. Hemodynamic parameters, such as blood pressure and heart rate, will be closely observed during the perioperative period to ensure patient safety.

Significance:

The findings from this study aim to identify a superior pain management strategy that minimizes opioid consumption, reduces side effects, and enhances recovery and patient satisfaction following MRM. If successful, the results could inform clinical practice and improve postoperative care for breast cancer patients.

This study is conducted at Ain Shams University hospitals and adheres to ethical guidelines to ensure the safety and well-being of all participants.

ELIGIBILITY:
Inclusion Criteria:

* Female patients older than 21 years old
* American Society of Anesthesiologists (ASA) physical status II.

Exclusion Criteria:

* Known allergy to one of the study's medications.
* Skin infections at the site of the needle puncture.
* Significant organ dysfunction (hepatic, renal, or cardiac dysfunction), coagulopathy or recent anticoagulant use, epilepsy.
* Patients diagnosed with obstructive sleep apnoea, pulmonary compromise .

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
Total amount of rescue pain medication required within the first 48 hours after surgery | 48 hours
  Researchers will report the total amount of analgesia used in the first 48 hours after surgery

SECONDARY OUTCOMES:
Time to first rescue analgesia' | 48 hours
  The time at which the first analgesia is adminstered after surgery
Total intraoperative fentanyl consumption | Total intraoperative time of surgery
  The total intraoperative consumption of fentanyl
Sleep quality | 48 hours
  The postoperative quality of sleep will be evaluated by The Pittsburgh Sleep Quality Index.
Time for the first ambulation | 48 hours
  The time at which the patient will be first be able to ambulate from bed.
VAS score for pain | 48 hours
  The postoperative pain using The Visual Analogue Scale (VAS) from 0 to 10, with two endpoints representing 0 ('no pain') and 10 ('pain as bad as it could be).
VAS score for nausea | 48 hours
  nausea during the postoperative period using Visual Analogue Scale (VAS) with two endpoints representing 0 ('no nausea') and 10 ('nausea as bad as it could be')
Patient Satisfaction score | 48 hours
  (five-point Likert scale) where (1 = extremely dissatisfied to 5 = extremely satisfied) to measure postoperative patient satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Ainshams University Hospitals, Cairo, Abbasiya, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaur U, Shamshery C, Agarwal A, Prakash N, Valiveru RC, Mishra P. Evaluation of postoperative pain in patients undergoing modified radical mastectomy with pectoralis or serratus-intercostal fascial plane blocks. Korean J Anesthesiol. 2020 Oct;73(5):425-433. doi: 10.4097/kja.20159. Epub 2020 Sep 24. PMID 32987492
- [Background] Hong B, Yoon SH, Youn AM, Kim BJ, Song S, Yoon Y. Thoracic interfascial nerve block for breast surgery in a pregnant woman: a case report. Korean J Anesthesiol. 2017 Apr;70(2):209-212. doi: 10.4097/kjae.2017.70.2.209. Epub 2017 Jan 12. PMID 28367293
- [Background] Zhang H, Miao Y, Qu Z. Refining a great idea: the consolidation of PECS I, PECS II and serratus blocks into a single thoracic fascial plane block, the SAP block-a concern on the muscle pain. Reg Anesth Pain Med. 2020 Jun;45(6):480. doi: 10.1136/rapm-2019-101042. Epub 2019 Oct 25. No abstract available. PMID 31653798
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Boogaerts JG, Vanacker E, Seidel L, Albert A, Bardiau FM. Assessment of postoperative nausea using a visual analogue scale. Acta Anaesthesiol Scand. 2000 Apr;44(4):470-4. doi: 10.1034/j.1399-6576.2000.440420.x. PMID 10757584